CLINICAL TRIAL: NCT00625261
Title: Effectiveness of a Parent-Based Language Intervention Group Program for Two-Year-Old Children With Language Delay
Brief Title: Effectiveness of Early Parent-Based Language Intervention
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Prof. Joachim Pietz, Department of Pediatric Neurology, Chidren´s Hospital, University of Heidelberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 243/2002
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Last update posted 2008-02-28 (Estimated); Status verified 2007-08

CONDITIONS: Language Delay; Developmental Language Disorders
Keywords: Language delay; Speech and language disorders; Early language intervention; Parent-based language intervention
MeSH Terms: conditions — Language Development Disorders; Speech; Language Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): The mothers of the two-years old children in the intervention group took part at the Heidelberg Parent-based Language Intervention HPLI
  Interventions: Other: Heidelberg Parent-based Language Intervention HPLI
- 2 (No Intervention): Waiting group, no intervention until children were three years of age

INTERVENTIONS:
Other: Heidelberg Parent-based Language Intervention HPLI — The HPLI is a group program for parents of young children with language delay. This 12-14week program includes seven two-our sessions and one three-our session six months later. It is designed for 5 to 10 people and based of an interactive model of language intervention, wich presumes that optimized parental input will provide better language-learning opportunities.
  Other Names: Early language intervention
  Arms: 1

SUMMARY:
The purpose of the study is to examine the effectiveness of a highly-structured parent-based language intervention group program for two-year-old children with language delay.

DETAILED DESCRIPTION:
Language delay in toddlers is a prevalent problem for pediatric practitioners. As there are no clear guidelines to deal with this problem, in German speaking countries the "wait-and-see"approach is widely chosen, although longitudinal studies have found that children with language delay are at risc for cognitive, behavioral and social-emotional problems.

During the last few years various forms of early language intervention have been increasingly implemented in German speaking countries. However, they have not been evaluated.

Early parent-based intervention could be an economical way in prevention speech and language disorders.

ELIGIBILITY:
Inclusion Criteria:

* Children with receptive and/or expressive language abilities below norm range measured by the standardized and norm-referenced German developmental language test SETK-2 (Grimm, 2000)

Exclusion Criteria:

* Children with visual impairments, genetic syndromes, metabolic diseases
* Children with previous language intervention

Ages: 24 Months to 27 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2003-10; Primary Completion 2008-02 (Actual); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Receptive and expressive language abilities using standardized instruments (SETK-2, SETK 3-5, AWST, HVS, HASE, HSET) | at 2; 6, 3, 4, 5 and 8 years of age

SECONDARY OUTCOMES:
Parent-report screening questionnaire ELFRA-2 (adoption of the MacArthur Communicative Development Inventories-CDI); cognitive and social-emotional development assessed by standardized instruments, | at 2;6, 3, 4, 5 and 8 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Anke Buschmann, MA, Principal Investigator — Department of Pediatric Neurology, Children´s Hospital, University of Heidelberg
Locations (1):
- Department of Pediatric Neurology, Childrens Hospital, University of Heidelberg, Heidelberg, Germany